CLINICAL TRIAL: NCT00170118
Title: Effects of Motivational Interviewing on Self-Efficacy and Standardized Low Back Pain Outcomes in Patients With Chronic Back Pain
Brief Title: Effects of Motivational Interviewing on Self-Efficacy and Standardized Low Back Pain Outcomes in Patients With Chronic Back Pain"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: 49-05
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2010-01-28 (Estimated); Status verified 2010-01

CONDITIONS: Chronic Low Back Pain
MeSH Terms: interventions — Motivational Interviewing

INTERVENTIONS:
Behavioral: motivational interviewing

SUMMARY:
The majority of the study consists of standard of care treatment for people with low back pain that has lasted more than three months. Half of the participants in the study will receive physical therapy from physical therapists that have received additional training in an educational technique. In order to determine if there is a difference in patient outcome when the educational technique is used, you will be asked to complete five short surveys before receiving physical therapy (10 minutes total). A sample of the physical therapy sessions using the educational technique will be videotaped. The videotape will be of the physical therapist to prove they did use the educational technique, not of you the participant in the study. You will remain anonymous and will not be used and the tape will not be used for publication or presentation purposes. You will also be asked to complete one survey after participating in physical therapy (2 minutes), and all five short surveys (10 minutes total) six weeks after your last physical therapy session.

You will be put in one of 2 groups by chance (as in the flip of a coin). A computerized selection process will be used to assign participants to the study. You will not know if you are in the study group or the non-study group.

DETAILED DESCRIPTION:
This is a pilot study to evaluate the impact of MI on self-efficacy and outcomes for chronic low back pain.

Design Prospective randomized, single blind pilot, controlled study. Patients will be referred from E10 and the Spine Center by contacting the study coordinator. The Coordinator will meet with potential participants, determine if they meet the inclusion and exclusion criteria, obtain informed consent, assess self-efficacy using the Stanford Self efficacy instrument, use en bloc randomization for self-efficacy to the experimental and control group. They will then complete the SF-12, a VAS pain scale, and the Roland and Morris Disability questionnaire, a few questions about employment status and 1 question about satisfaction with care.

The experimental group(goal n=20) will be treated by physical therapists that have been trained in motivational interviewing techniques by a PhD and a sample of these sessions will be videotaped for validation purposes. The control group(goal n=20) will receive PT from any PT as per the normal standard of care.

Both the experimental and control group will complete an additional self-efficacy instrument prior to leaving. Six weeks after the patients participate in a motivational interview session they will be mailed a repeat of all of the previously mentioned instruments including the self-efficacy tool. Patients who return the completed instruments will receive forty dollars. If effect size is small, this pilot study will be underpowered, if a clinically significant trend is observed additional funding will be sought and the experimental and control n will be expanded to 64.

Setting Tertiary academic medical center Participants Referrals from a Spine Center, or a large outpatient Physical Medicine and Rehabilitation practice with at least three months of chronic low back pain.

Primary Outcome Measure Self-efficacy for Managing Chronic disease 6-Item scale

Main Outcome Measures Roland and Morris Disability Questionnaire Pain VAS Satisfaction with care question Disability status question SF-12 Exclusion Criteria Medical /legal involvement Active workers compensation Infection or tumor in spine Active systemic disease in the lumbar spine Multiple other musculoskeletal problems that require Treatment Patients receiving more than 2 PT sessions

Inclusion Criteria Three or more months of low back pain Ability to read, write and speak English

ELIGIBILITY:
Exclusion Criteria Medical /legal involvement Active workers compensation Infection or tumor in spine Active systemic disease in the lumbar spine Multiple other musculoskeletal problems that require Treatment Patients receiving more than 2 PT sessions

Inclusion Criteria Three or more months of low back pain Ability to read, write and speak English

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2005-06; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
SF - 12
Self-efficacy for Managing Chronic disease 6-Item scale
Roland and Morris Disability Questionnaire
Pain Visual analog scale
Satisfaction with care question

SECONDARY OUTCOMES:
Disability status question

CONTACTS AND LOCATIONS:
Overall Officials: Catherine K. Schmidt, MS DO, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States